CLINICAL TRIAL: NCT04818333
Title: Phase I/II Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-A1811 for Injection in Subjects With Advanced Non-small Cell Lung Cancer Who Have HER2 Expression , Amplification, or Mutation
Brief Title: A Study of SHR-A1811 in Subjects With Advanced Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-I-103
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Intervention Model Description: Single arm study of SHR-A1811
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental): SHR-A1811 was administered intravenously every 3 weeks (Q3W) until discontinuation treatment
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — Phase 1 Drug: SHR-A1811 There are four pre-defined dose regimens . Subjects will be enrolled with an initial dose Phase 2 Drug: SHR-A1811 Doses will be determined from Phase 1

SUMMARY:
This is an open-label, two-part study to evaluate the safety, tolerability, pharmacokinetics, and efficacy of SHR-A1811 for injection in subjects with advanced non-small cell lung cancer who have HER2 expression , amplification, or mutation

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. advanced non-small cell lung cancer with HER2 expression , amplification, or mutation
4. has previously received platinum-based chemotherapy for advanced or metastatic NSCLC, has developed disease progression during or after treatment, or is unable to tolerate platinum-based chemotherapy.
5. There is at least one measurable lesion according to RECIST V1.1 criteria

Exclusion Criteria:

1. Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0 grade ≤ 1.
2. Has received HER2 antibody drug conjugates,
3. Central nervous system metastasis or meningeal metastasis with clinical symptoms
4. Has active infection requiring systemic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1:Incidence of Adverse Events (AEs) by CTCAE v5.0 of SHR-A1811 | From Day 1 to90 days after last dose ，appropriately to 3 years
  Assess safety and tolerability of SHR-A1811 by way of adverse events (CTCAE v5.0)
Phase 1:Severity of Adverse Events (AEs) by CTCAE v5.0 of SHR-A1811 | From Day 1 to90 days after last dose ，appropriately to 3 years
  Assess safety and tolerability of SHR-A1811 by way of adverse events (CTCAE v5.0)
Phase1: Maximum tolerated dose (MTD) | 12 months
  Incidence rate and category of dose limiting toxicities (DLTs) during the first 21-day cycle of SHR-A1811 treatment
Phase 1: Recommended Phase 2 dose (RP2D) | 12 months
  RP2D was determined based on the safety, tolerability, PK, immunogenicity data and efficacy information obtained
Phase2:ObjectiveResponse Rate (ORR) | Subjects were evaluated on tumor imaging every 6 weeks after treatment initiation and every 12 weeks after 54 weeks, until imaging progression, initiation of new antitumor therapy, loss of follow-up, and death，appropriately to 3 years
  As assessed by RECIST v1.1 , as assessed by independent review committee (IRC)

SECONDARY OUTCOMES:
Phase 1：PK parameter ：Tmax of SHRA1811 | appropriately to 3 years
  Time to maximal concentration (Tmax) of SHR-A1811
Phase1:PK parameter: Cmax of SHR-A1811 | appropriately to 3 years
  Maximal concentration (Cmax) of SHR-A1811
Phase1:PK parameter: AUC0-t of SHR-A1811 | appropriately to 3 years
  AUC computed from time zero to the time of the last quantifiable concentration (AUC0-t) of SHR-A1811
Phase1:Immunogenicity of SHR-A1811 | Immunogenicity sample collection time points include: within 30 min before administration of C1D1, C2D1, C3D1, C4D1, C6D1 and C8D1 starting from cycle 11 only in every 3 cycles ,appropriately to 3 years
  Including anti-drug antibody and/or neutralizing antibody
Phase2:Progression Free Survival (PFS) | appropriately to 3 years
  As assessed by RECIST v1.1 , as assessed by independent review committee (IRC) and investigator
Phase2:ObjectiveResponse Rate (ORR) | appropriately to 3 years
  As assessed by RECIST v1.1 , as assessed by investigator
Phase2:Duration of response (DOR) | appropriately to 3 years
  As assessed by RECIST v1.1 , as assessed by independent review committee (IRC) and investigator
Phase2:Disease control rate (DCR) | appropriately to 3 years
  As assessed by RECIST v1.1 , as assessed by independent review committee (IRC) and investigator
Phase2:Overall survival (OS) | Approximately 5 years after last subject enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li Z, Wang Y, Sun Y, Wang L, Li X, Sun L, He Z, Yang H, Wang Y, Wang Q, Song Z, Hong W, Wang Y, Xia G, Yu Y, Peng M, Song Y, Wang D, Meng R, Fang J, Luo Y, Liang W, Hu S, Wang Z, Song K, Li Y, Yang L, Shi W, Lu S. Trastuzumab rezetecan, a HER2-directed antibody-drug conjugate, in patients with advanced HER2-mutant non-small-cell lung cancer (HORIZON-Lung): phase 2 results from a multicentre, single-arm study. Lancet Oncol. 2025 Apr;26(4):437-446. doi: 10.1016/S1470-2045(25)00012-9. Epub 2025 Feb 25. PMID 40020696
- [Derived] Li Z, Song Z, Hong W, Yang N, Wang Y, Jian H, Liang Z, Hu S, Peng M, Yu Y, Wang Y, Jiao Z, Zhao K, Song K, Li Y, Shi W, Lu S. SHR-A1811 (antibody-drug conjugate) in advanced HER2-mutant non-small cell lung cancer: a multicenter, open-label, phase 1/2 study. Signal Transduct Target Ther. 2024 Jul 15;9(1):182. doi: 10.1038/s41392-024-01897-y. PMID 39004647